CLINICAL TRIAL: NCT00053469
Title: Early Learning and Development Project
Brief Title: Infant s Examination and Manipulation of Objects
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030069; 03-CH-0069
Record Dates: First submitted 2003-01-30; First posted 2003-01-30 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-03-30

CONDITIONS: Healthy; Infant
Keywords: Cognitive Development; Motor Planning; Categorization; Perception; Adaptation

SUMMARY:
This study will explore how babies become able to use their experience with objects to plan to manipulate them appropriately. For example, an adult knows that picking up a grocery bag full of canned food requires different actions than are needed for lifting an empty bag. This study will examine when and how infants first begin to adapt their actions to manipulate specific objects that weigh different amounts.

Participants will include normal healthy babies within 2 weeks of their first birthday. If the expected results are obtained from testing, 9-month-old children will then be studied to identify a lower age boundary in task performance. If the expected results are not obtained at the 12-month test age, older children will be recruited to participate.

The study involves one 30-minute session with the baby and his or her mother or father. The parent will answer some questions about the family, such as its size and ethnic make-up. The infant will then have small magnetic sensors taped to the underside of each arm and to the back. While sitting on the parent s lap, the infant will be presented with plastic toys, and his or her actions will be measured by the sensors as he or she reaches for and picks up the toys. The sensors will be connected to a computer that will track and record the motion of the infant s arms.

...

DETAILED DESCRIPTION:
The major objective of this research is to better understand the functional significance of object categorization in early development. The proposed work is designed to examine the emergence of infants ability to access internal categorical representations in service of planning actions on the external environment. Representation, in this capacity, refers simply to stored information that can influence later behavior. Categorization refers to the treatment of discriminable objects as equivalent in some way. Even very young infants appear able to visually categorize diverse sets of discriminable patterns or objects, and can form internal representations of such bounded collections. Much less is known, however, about infants ability to actually utilize such representations in the guidance of goal directed action. The present research is designed to characterize the functional and behavioral significance of object representations in infancy, focusing particularly on categorically organized representations. The primary research strategy to be used consists of analyzing infants examination and manipulation of novel objects that vary both in visual (i.e., shape and color) as well as nonvisual dimensions (i.e., weight). In a laboratory procedure, twelve-month old infants will explore novel objects of different weights, and their subsequent handling of modified test objects will be measured with an electronic motion analysis system. Kinematic analyses of infants actions on the test objects will reveal how these actions were prepared in relation to their previous experience with similar objects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Infants will be selected for inclusion in each study on the basis of age, gestational status (i.e., full-term vs. pre-term birth), visual normality, and general health status.

The initial group will be recruited to participate within two weeks on either side of their first birthday (12 months of age).

Equal numbers of males and females will be recruited to participate. If the sample participating in either experiment fails to perform in the manner expected, additional participants will be recruited at older test ages to identify when in the course of development such behavioral guidance emerges. As successive test ages will be separated by 6 month intervals, independent samples of 18-, then 24-month-old children will be recruited until the expected pattern of adaptive actions is observed (cf. Fossberg, et al., 1992).

EXCLUSION CRITERIA:

Infants with a gestational age of less than 36 weeks, and/or those with histories of severe perinatal complications, visual abnormalities, or congenital developmental disorders will not be recruited for participation.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2003-01-28; Study Completion 2015-03-30

CONTACTS AND LOCATIONS:
Overall Officials: Clay W. Mash, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adolph KE. Learning in the development of infant locomotion. Monogr Soc Res Child Dev. 1997;62(3):I-VI, 1-158. PMID 9394468
- [Background] Baillargeon R. Representing the existence and the location of hidden objects: object permanence in 6- and 8-month-old infants. Cognition. 1986 Jun;23(1):21-41. doi: 10.1016/0010-0277(86)90052-1. No abstract available. PMID 3742989
- [Background] Bornstein MH, Kessen W, Weiskopf S. Color vision and hue categorization in young human infants. J Exp Psychol Hum Percept Perform. 1976 Feb;2(1):115-29. doi: 10.1037//0096-1523.2.1.115. PMID 1262792